CLINICAL TRIAL: NCT00556855
Title: A 4-Week Randomized, Double-Blind, Placebo-Controlled, Right-Left Comparison Study With E-DO in Chronic Hand Dermatitis
Brief Title: Comparison Study With E-DO in Chronic Hand Dermatitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HenKan Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Joseph Tseng, HenKan Pharmaceutical Co., Ltd.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EDO-CHD001
Record Dates: First submitted 2007-11-08; First posted 2007-11-12 (Estimated); Last update posted 2009-01-12 (Estimated); Status verified 2009-01

CONDITIONS: Chronic Hand Dermatitis
Keywords: chronic hand dermatitis; research study; E-do; HK-03

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental): applied on one hand
  Interventions: Other: E-DO
- B (Placebo Comparator): applied on the other hand
  Interventions: Other: Placebo

INTERVENTIONS:
Other: E-DO — topical lotion, once daily (evening), total duration: 4 weeks
  Other Names: HK-03
  Arms: A
Other: Placebo — topical lotion, once daily (evening), total duration: 4 weeks
  Other Names: Vehicle
  Arms: B

SUMMARY:
The objective of this study is to evaluate the topical E-DO in patients with Chronic Hand Dermatitis (fu kuei shou).

DETAILED DESCRIPTION:
Hand dermatitis, also called fu kuei shou, is a skin condition in which the hands develop a rash and become red, dry, cracked, and inflamed. This is a very common occuring in about 10% of women and 4% of men. The condition can eventually cause pain on contact with even simple solutions such as water. Hand dermatitis is particularly common in industries involving cleaning, catering, metalwork, hairdressing, healthcare and mechanical work, and is often difficult to be treated effectively. Some patients develop varying levels of disability due to lack of acceptable effective treatments and may be forced to change occupations in order to achieve relief.

Primary treatment for hand dermatitis is typically topical corticosteroids, especially when the offending agent(s) cannot be identified or avoided. However, patients may eventually develop tachyphylaxis to the anti-inflammatory activity of mid-potency or high-potency topical corticosteroids and patients with severe, chronic involvement may often be less likely to respond. Potential topical alternatives to corticosteroids include psoralen plus ultraviolet (PUVA), but the phototherapies are inconvenient because multiple clinical visits are required and hand phototherapy units may not be available.

Moisturizers have been found to help restore the skin barrier providing a protective layer on surface of the skin to trap water and prevent the penetration of irritants and allergens. An emollient cream is superior in trapping the moisture within the skin. Emollients may form a covering film, which acts as a barrier for chemicals from the exterior and which restricts the loss of water and other essential substances from the interior. E-DO gel is a potential agent for revitalizing our skin cells so that regain their moisture retention capacity.

E-DO has known significant improvements in wound healing and the inhibition of Staphylococcus aureus and Propionibacterium acnes. This pilot research trial will investigate the effect of topical E-DO for patients with hand dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Males or females aged 20 years of age or above;
* Patients must have chronic hand dermatitis based upon clinical diagnosis at least mild dermatitis of the both hands at baseline, as defined by an Investigator Global Assessment score of 2 (mild) to 5 (very severe);
* Patients must have been informed of the study procedures and therapies and have given their written informed consent.

Exclusion Criteria:

* Women who are pregnant or who are breast-feeding;
* Patients who have received systemic corticosteroids (i.e., oral, intravenous, intra-articular, rectal, intramuscular) within one month prior to first application of study medication;
* Patients who have received phototherapy (e.g., UVB, PUVA) or systemic therapy (e.g., immunosuppressants, cytostatics) known or suspected to have an effect on hand dermatitis within one month prior to first application of study medication;
* Patients who are treated with topical therapy (e.g., tar, topical corticosteroids) known or suspected to have an effect on hand dermatitis within 7 days prior to first application of study medication;
* Patients who have a diagnosis on the hands of active atopic dermatitis, dyshidrotic eczema, psoriasis, urticaria, active fungal or bacterial infection, or identified allergic contact dermatitis (e.g., poison ivy dermatitis)
* Patients with hypersensitivity to vitamin B, vitamin C, vitamin E, beta-carotene.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2007-12; Primary Completion 2008-07 (Actual); Study Completion 2008-07 (Actual)

PRIMARY OUTCOMES:
The therapeutic response rate (clear or almost clear) base on Investigator Global Assessment (IGA) | at Week 4 (or at time of early discontinuation)

SECONDARY OUTCOMES:
The proportion of the patients with at least 50% improvement (clinically significant response) base on the patient's global assessment (PaGA) | at Week 4 (or at time of early discontinuation)
The percent change in the HEAS (Hand Eczema Area and Severity Score) from baseline to post-treatment. | during 4 Weeks
The change of pruritus score and pain score from baseline to post-treatment | during 4 weeks
The change in the degree of moisture on the skin's surface, and the water evaporation on skin surfaces by TEWL, and the QOL scores from baseline to the end of study. | End of study (4 weeks)
The safety and tolerability of E-DO including AE/SAE report | during 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Chia-Yu Chu, MD, PhD, Principal Investigator — Department of Dermatology, Nation Taiwan University Hopital, R.O.C.
Locations (1):
- Department of Dermatology, NTUH, Taipei, Taiwan